CLINICAL TRIAL: NCT00557011
Title: A Phase 2, Randomized, Double-Blind, Placebo- and Active-Controlled, 3-Treatment, 3-Period, Crossover Study With One Week Per Treatment and Once-a-Day Dosing of Either NRP104, Adderall XR, or Placebo in Children Aged 6 to 12 Years With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: NRP104, Adderall XR or Placebo in Children Aged 6-12 Years With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New River Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRP104.201
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; SLI381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): NRP104
  Interventions: Drug: NRP104
- 2 (Active Comparator): Adderall XR
  Interventions: Drug: Adderall XR
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NRP104 — 30 mg, 50 mg or 70 mg capsules taken orally once daily in the morning
  Other Names: lisdexamfetamine dimesylate
  Arms: 1
Drug: Adderall XR — 10 mg capsules taken once daily in the morning at dosages of either 1x10mg, 2x10mg or 3x10mg
  Other Names: mixed salts of a single-entity amphetamine
  Arms: 2
Drug: Placebo — Placebo capsule taken once daily in the morning
  Arms: 3

SUMMARY:
The purpose of this study is to assess, in a controlled environment, the efficacy and safety of NRP104 and Adderall XR compared to placebo in treatment of children, aged 6-12, with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* males and non-pregnant females, aged 6-12 years DSM-IV-TR criteria for diagnosis of ADHD, combined or hyperactive-impulsive subtypes
* on stable regimen of stimulants for at least one month in the last six months and has shown adequate response to stimulants without unacceptable side effects

Exclusion Criteria:

* co-morbid psychiatric diagnosis such as psychosis, bipolar illness, severe OCD, severe depressive or anxiety disorder
* history of seizure during the last 2 years, a tic disorder or Tourette's
* clinically significant ECG or laboratory abnormalities at screening or baseline
* taking clonidine or anticonvulsant drugs
* taking medications that affect blood pressure or heart rate

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2004-09; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
SKAMP-DS scores across a treatment assessment day | 1 week

SECONDARY OUTCOMES:
SKAMP Attention Scale, PERMP attempted score, PERMP correct score, and CGI scores across the treatment assessment day | 1 week
Treatment emergent adverse events | 1 week
PK profile and PK/PD relationship of NRP104 | After multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, M.D., Principal Investigator — Harvard Medical School (HMS and HSDM); Samuel Boellner, M.D., Principal Investigator — Clinical Study Centers, LLC; Ann Childress, M.D., Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.; Frank Lopez, M.D., Principal Investigator

REFERENCES:
- [Result] Biederman J, Boellner SW, Childress A, Lopez FA, Krishnan S, Zhang Y. Lisdexamfetamine dimesylate and mixed amphetamine salts extended-release in children with ADHD: a double-blind, placebo-controlled, crossover analog classroom study. Biol Psychiatry. 2007 Nov 1;62(9):970-6. doi: 10.1016/j.biopsych.2007.04.015. Epub 2007 Jul 12. PMID 17631866
- [Derived] Faraone SV, Spencer TJ, Kollins SH, Glatt SJ. Effects of lisdexamfetamine dimesylate treatment for ADHD on growth. J Am Acad Child Adolesc Psychiatry. 2010 Jan;49(1):24-32. doi: 10.1097/00004583-201001000-00006. PMID 20215923
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html